CLINICAL TRIAL: NCT06099106
Title: Evaluation of the Safety and Performance of ENDOMATIC SEPIOLA Left Atrial Appendage (LAA) Closure Device in Patients With Atrial Fibrillation
Brief Title: Safety and Performance of ENDOMATIC SEPIOLA Left Atrial Appendage (LAA) Closure Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endomatic Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS-6283
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantable device (Experimental): Endomatic SEPIOLA System
  Interventions: Device: SEPIOLA System

INTERVENTIONS:
Device: SEPIOLA System — Implantation of the SEPIOLA device into the left atrial appendage.

SUMMARY:
The study is designed to evaluate the safety and performance of the ENDOMATIC SEPIOLA Left Atrial Appendage (LAA) Closure Device in Patients with non-valvular Atrial Fibrillation, who are at increased risk for stroke, and that cannot take, or have a reason to seek an alternative, to long-term anticoagulation therapy.

Potential patients who are candidates for LAA closure will be screened to confirm that all inclusion/exclusion criteria are met, with final eligibility confirmation on day of procedure.

All enrolled subjects who went through the procedure will be followed during the procedure to hospital discharge.

Additional follow up time points are scheduled at 45 days, 6 months and 12 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* calculated CHA2DS2-VASc score of 2 or greater.
* The subject is non-eligible or have an appropriate rationale to seek a non-pharmacologic alternative to chronic oral anticoagulants.
* documented non-valvular atrial fibrillation
* Subject suitable for vascular/cardiac intervention procedure
* suitable LAA anatomical measurements for study device

Exclusion Criteria:

* Subject who requires anticoagulation for a condition other than AF.
* NYHA classification IV.
* Complex congenital heart disease.
* Presence of circumflex coronary artery stent.
* The subject has a prosthetic valve in any position.
* atrial septal defect closure or has an ASD/PFO device.
* presence of intracardiac thrombus.
* Any cardiac surgery in the past
* LVEF < 35%.
* intracardiac thrombus
* moderate or severe mitral valve stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
SEPIOLA System Safety | 7 days, 45 days and 6 months post procedure
  Device and Investigational Procedure Related Serious Adverse Events (SAE)

SECONDARY OUTCOMES:
Device success | 45 days
  Confirmation of functional LAA closure

CONTACTS AND LOCATIONS:
Locations (5):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
- Vilnius university hospital Santaros Klinikos, Vilnius, Lithuania
- Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan, Poland
- Ezgu Niyat, Tashkent, Uzbekistan